CLINICAL TRIAL: NCT01693965
Title: Clinical Course and Changes in the Respiratory Microbiota Based on Antibiotic Treatment in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-A00601-42; 2012-14 (Other: AP HM)
Record Dates: First submitted 2012-09-13; First posted 2012-09-26 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Bronchopulmonary Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sputum samples (Other)
  Interventions: Other: sputum samples

INTERVENTIONS:
Other: sputum samples

SUMMARY:
Bronchopulmonary infection is the most common and serious complication in the evolutionary course of cystic fibrosis (CF). Administration of antibiotics adapted to infecting pathogens is one of the key issues for its management. However, more than half of patients with CF have chronic respiratory infections for which infectious agent remains unknown leading to empirical antibiotic therapies that are not adapted to the causative agents. Recently, new technologies have been applied for the description and characterization of microbial agents in CF patients including molecular biology techniques that allowed us to detect and to identify new and/or emerging pathogens. Moreover, more sophisticated molecular techniques such as pyrosequencing and PCR amplification and cloning lead us to demonstrate the huge microbial diversity associated with chronic bronchopulmonary infections in this population. Otherwise, a metagenomic approach revealed the extraordinary complexity of the respiratory flora in these patients and, somewhat unexpected, abundance of anaerobes, viruses, and bacteriophages. In addition, it has been shown that some antibiotics commonly used in clinical practice for the treatment of respiratory infections were able to induce these bacteriophages, suggesting the existence of lateral gene transfer by transduction. The human microbiome is the set of microbial communities associated with the human body and represents all living microorganisms in the body. Its role in the immunity development has recently been demonstrated suggesting that changes in this ecosystem play a critical role in evolution of several human diseases. For example, in obesity it has been shown that there is a relationship between the intestinal human microbiota and nutritional and metabolic status of the hosts and specific alterations of these intestinal microbiota may represent a metagenomic signature of this disease. Evolution of the respiratory microbiota in patients with cystic fibrosis, whose nutritional status is often impaired (chronic malnutrition due to disorder of digestive absorption) and receiving regular antibiotic treatments remains unknown to date. Characterization of this ecosystem and its role is a critical step to understand the evolutionary course of the disease.

The main objective of this seminal study is to describe and to characterize the respiratory microbiota from sputum samples obtained from a limited number of selected patients with CF from 5 regional care centers (CRCM) from South of France (Mucomed network) (2 patients per center : 6 adults and 4 children), with similar clinical, microbiological and functional status before and after a cure of antibiotics. Different microbiological tools will be used including axenic culture systems, co-culture on amoebae in order to to isolate and to identify the microbial communities. Identification of bacteria will be done using MALDI-TOF mass spectrometry and/or molecular techniques. Moreover, 16S rRNA PCR amplification followed by cloning and sequencing of PCR products from the same sputum sample will be carried out to identify and to compare the bacterial species identified using molecular methods. In a second step, once the respiratory microbiota was characterized, it will be interesting to develop a dedicated microarray that will allow to detect all the bacteria identified in the first stage of the project and to assess its relevance on a larger cohort of patients with CF by studying the correlation between the respiratory microbiota and clinical status of patients according to the prescribed antibiotic treatments.

This study will open new clinical perspectives and will help us to determine the potential role of antibiotics on the microbiota evolution during treatment according to regional health care practices. This will contribute to better understand the role of the microbiota in the evolution of these chronic respiratory infections. It could be the first step for innovative therapeutic strategies, taking into account the balance of complex microbial flora and possibly evolving according to antibiotic therapies. It could also form part of a larger preventive strategy against transmission of specific pathogens in CF.

ELIGIBILITY:
Inclusion Criteria:

* Subjects achieves of cystic fibrosis followed regularly in one 5 Grown-up CRCM or Children involved in the study

  * Inclusions of 10 patients at the rate of 2 subjects by center (6 adults and 4 children). The adults (> 18 years) will be patients followed in the CRCM of grown-up Marseille (2), of Giens-Hyères (1), Montpelier (1) and Nice (2); 4 children ( 11 - 17 years) will be followed in the CRCM of Marseille children (2), of Giens-Hyères (1) and Montpelier (1).
  * Patients having a clinical status (appeal(recourse) to 1 cure / year of antibiotics in IV), functional (VEMS = 30 % of the theoretical value) and microbiological identical,
  * Patients presenting a bronchial colonization to Pseudomonas aeruginosa known for at least 3 months, sensitive to the tobramycine and to the ceftazidime, not having received from cure of antibiotic IV during month preceding the inclusion in the study.
  * Patients not presenting fungal concommitante colonization or for at least 3 months

Exclusion Criteria:

* not affected Subject of cystic fibrosis

  * Subject achieves of cystic fibrosis followed regularly in another center than the one 4 participating CRCM
  * Subject achieves of cystic fibrosis among which the clinical status and the initial bronchial colonization is not known
  * Subject having meant in the oral its opposition has the study

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
A taking of expectorations | 3 years
  describe and characterize the respiratory microbiota

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France